CLINICAL TRIAL: NCT07275125
Title: Outcomes of Drug Resistant Epileptic Pediatric Patient by Modified Atkins Diet
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Saber Elsayed, Resident, Sohag University
Other Study IDs: Soh-med-25-9-IMS
Record Dates: First submitted 2025-09-28; First posted 2025-12-10 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-11

CONDITIONS: Drug Resistant Epilepsy
MeSH Terms: conditions — Drug Resistant Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To assess clinical outcomes in drug resistant epileptic pediatric patient by modified atkin diet with focusing on following points:

1. Control of seizures(frequency , duration and numbers of hospital admissions) .
2. Quality of life by pediatric quality of life inventory v4.
3. Cognitive function by stanford binet intelligence scale 5th edition.
4. Growth parameters ( weight, height will be combined to report BMI in kg/m^2).

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1-18 years.
* Diagnosed with drug-resistant epilepsy according to ILAE definition.[2]
* On KD for at least 6 months.

Exclusion Criteria:

* - Patients with contraindicated metabolic/genetic conditions.
* Non-compliance with KD .

Patients on alternative dietary therapies (e.g., low glycemic diet)

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: This study will include pediatric patients with drug-resistant epilepsy (DRE) attending the ketogenic diet clinic at the Pediatric Neurology Unit, Sohag University Hospital. Eligible participants are children aged 1-18 years who meet the International League Against Epilepsy (ILAE) definition of DRE and have been on a ketogenic dietary therapy, specifically the Modified Atkins Diet (MAD), for at least 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
1-Control of seizures(frequency and duration of seizures) . 2-Quality of life by pediatric quality of life inventory v4. 3-Cognitive function by stanford binet intelligence scale 5th edition. 4-Growth parameters (weight and height by BMI in kg/m^2) | 6 month

SECONDARY OUTCOMES:
to detect clinical predictors of seizures control ( frequency of attack and duration) in patients with drug resistant epilepsy using MAD. | 6 month

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag faculty of medicine, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided